CLINICAL TRIAL: NCT03465943
Title: Crystalloid Versus Crystalloid and Colloid Combination Preload for Prevention of Hypotension in Patients Undergoing Elective Caesarean Section Under Intrathecal Anesthesia
Brief Title: Different Preloads for Prevention of Hypotension in Patients Undergoing Elective CS Under Intrathecal Anesthesia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rafeek Ramez Shawky Aziz, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Hypotension in elective CS
Record Dates: First submitted 2018-03-03; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Hypotension Drug-Induced
MeSH Terms: conditions — Hypotension | interventions — Crystalloid Solutions; HES 130-0.4

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ringer (Active Comparator): This group will receive 1 L of Ringer's solution as a preload
  Interventions: Drug: Ringer
- Voluven (Active Comparator): This group will receive 500 ml of 6% hydroxyethyl starch ( Voluven ) and 500 ml Ringer's solution as a preload
  Interventions: Drug: Ringer; Drug: Voluven

INTERVENTIONS:
Drug: Ringer — 1L of Ringer's solution as a preload in one group.
  Other Names: Crystalloid
Drug: Voluven — 500 ml of voluven will be given in combination with 500 ml Ringer's solution as a preload in the other group.
  Other Names: Hydroxyethyl starch 6%
  Arms: Voluven

SUMMARY:
The aim of this study was to compare between crystalloid versus crystalloid and colloid combination preloads for prevention of hypotension following intrathecal anaesthesia in patients undergoing elective Caesarean section.

To examine weather baseline perfusion index could predict the incidence of intrathecal-induced hypotension during Caesarean section.

DETAILED DESCRIPTION:
Intrathecal anesthesia is the most commonly used technique for elective Caesarean section all over the world.

One of the most common complications of this technique is hypotension. It's incidence is more than 80% without any prophylactic measures, this hypotension has adverse effects on both mother ( causing nausea and vomiting ) and foetus ( causing acidosis and neurological defects ).

This complication can be managed by several ways like fluid therapy, usage of vasopressors or combination between both of them.

Among the type of fluids ( crystalloid or colloid ) it's still not known which one of them is better. Crystalloid has a short intravascular half-life because of its rapid distribution into the interstitial space. On the other hand colloid remains longer within the intravascular space.

Change in baseline peripheral vascular tone due to pregnancy may affect the degree of such hypotension. The perfusion index ( PI ) derived from a pulse oximeter has been used for assessing peripheral perfusion dynamics due to changes in peripheral vascular tone.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18-40 years
* ASA 1&2

Exclusion Criteria:

* Patients with morbid obesity.
* Pre-existing or pregnancy-induced hypertension.
* Known cardiovascular or cerebrovascular disease.
* Abnormal CTG tracing.
* Any other contraindications for intrathecal anaesthesia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypotension | 1 hour
  Decrease in systolic blood pressure more than 20% of base line

SECONDARY OUTCOMES:
Perfusion index | 1 hour
  Derived from pulse oximeter
Heart rate | 1 hour
Urine output | 1 hour

REFERENCES:
- [Background] Ripolles Melchor J, Espinosa A, Martinez Hurtado E, Casans Frances R, Navarro Perez R, Abad Gurumeta A, Calvo Vecino JM. Colloids versus crystalloids in the prevention of hypotension induced by spinal anesthesia in elective cesarean section. A systematic review and meta-analysis. Minerva Anestesiol. 2015 Sep;81(9):1019-30. Epub 2014 Dec 11. PMID 25501602
- [Result] Ngan Kee WD. Confidential enquiries into maternal deaths: 50 years of closing the loop. Br J Anaesth. 2005 Apr;94(4):413-6. doi: 10.1093/bja/aei069. No abstract available. PMID 15758080